CLINICAL TRIAL: NCT02970994
Title: Linear Growth and Neurobehavioural Outcome in Preterm Neonates (<34 Weeks) at 37 Weeks and 40 Weeks of Corrected Gestational Age : a Prospective Observational Study
Brief Title: Linear Growth and Neurobehavioural Outcome in PT Neonates (<34 Wks) at 37 and 40 Wks of CGA
Status: Completed | Type: Observational
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, DR. VIKRAM DATTA, Professor, Lady Hardinge Medical College
Other Study IDs: LadyHardinge MC
Record Dates: First submitted 2016-11-12; First posted 2016-11-22 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: PreTerm Birth
Keywords: Linear growth and neurodevelopment outcome; < 34 weeks
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Preterm neonates <34 wks: Haemodynamicaly stable preterm neonates <34 weeks with in 48 hours of admission

SUMMARY:
This study will evaluate the association of linear growth on neurobehavioural outcome in preterm neonates at 37 and 40 weeks of (CGA) corrected gestational age.

DETAILED DESCRIPTION:
Growth of the preterm infant has historically been defined as weight gain over time. As weight gain and nutrition have been more extensively studied and their relationships with neurodevelopmental outcomes have been established, other growth parameters and their relationships to outcome need to be assessed.

Large multicenteric studies have demonstrated that poor postnatal weight gain has a negative effect on neurodevelopment . However, the neurodevelopmental consequences of linear stunting in this population were not assessed .Understanding this relationship is important because organ growth and differentiation are more closely linked to lean body mass and thus linear growth than to weight gain or fat mass alone. Moreover, weight gain and linear growth are not always tightly linked and may be influenced by both nutritional and non nutritional factors.

Linear growth represents lean body mass and protein accretion and also indexes organ growth and development, including the brain. American Academy of Pediatrics (AAP) recommends that preterm infants should grow similar to the fetus,but this guideline has been mostly applied to weight gain. As already described, the ideal weight gain to optimize neurodevelopmental outcomes has been studied extensively. However, ideal linear growth has yet to be defined. Intrauterine linear-growth velocity is approximately 1 cm/wk,and therefore is the goal that most neonatologists currently follow.Given the increasing evidence that linear-growth suppression is associated with poorer cognitive outcomes,length may now be an important anthropometric biomarker for later neurodevelopment. Research is needed to determine optimal goals of linear growth for preterm infants so as to optimize later growth and neurodevelopmental outcomes.

Recently the role of neurobehaviour has evaluated as early as at 37-40 weeks of CGA and is being predicted as an useful adjunct to the 12-18 month full neurodevelopmental assessment .Neurobehavioural assessment by tools like NAPI have been shown to correlate with BSID score at 18 months of corrected gestational age in preterm neonates.This has tremendous implications in terms of initiating an early rehabilitation /stimulation program for these neonates..

There is insufficient data on Correlation of linear growth and neurological outcome in preterm VLBW babies in India.With majority of VLBW neonates in India being SGA this assumes critical significance as growth faltering is reported to continue as late as 24 months postnatally.The linkage of linear growth faltering and poor neurodevelopmental outcome needs to be detected early in the India population and corrective strategies need to be instituted

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ( Haemodynamicaly stable preterm neonates <34 weeks with in 48 hours of admission )
* Parental Consent

Exclusion Criteria:

* Major congenital malformation
* Haemodynamic instability
* Birth asphyxia(Apgar score of less than 7 at 1 minute of age)
* Multiple gestation.
* IVH
* Meningitis
* Hypoglycemia at admission

Ages: 1 Day to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Haemodynamicaly stable preterm neonates <34 weeks with in 48 hours of admission
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Association of linear growth on neurobehavioural outcome in preterm neonates | 18 months
  All preterm neonates born in LHMC who meet the inclusion criteria will be included in the study with in 48 hours of admission .Demographic data, maternal history, labour details and neonatal details will be recorded in the proforma. Length will be measured using a flexible tape measuring tape and a standard infant length board to the nearest 0.1 cm . Length will be measured at time of enrolment,at time of discharge,at 37 weeks and 40 weeks of corrected gestational age.Standardized Z-scores will be calculated for the length and using reference data which included Fenton curves at birth and hospital discharge. Neonates will be evaluated by NAPI score at 37 weeks and 40 weeks of corrected gestational age for neurobehavioural assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Datta, MD,DNB, Principal Investigator — Lady Hardinge Medical College,New Delhi,Delhi,INDIA,110001.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pfister KM, Ramel SE. Linear growth and neurodevelopmental outcomes. Clin Perinatol. 2014 Jun;41(2):309-21. doi: 10.1016/j.clp.2014.02.004. Epub 2014 Apr 14. PMID 24873834